CLINICAL TRIAL: NCT07032363
Title: Implementing Depression and Adherence Treatment in HIV Care
Brief Title: Implementing Depression and Adherence Treatment
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: unclear reasons as to why the federal government is targeting grants with foreign components and putting them on hold unfairly and unethically
Sponsor: University of Miami (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven Safren, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20241034; R01MH136972 (NIH)
Record Dates: First submitted 2025-06-19; First posted 2025-06-24 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Depression; HIV; Adherence, Treatment; AIDS
Keywords: implementation science; HIV; depression
MeSH Terms: conditions — Depression; Treatment Adherence and Compliance; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Core (Other): Clinics in this arm will receive strategies that involve capacity building for nurses and education on mental health.
  Interventions: Other: Core Implementation Strategies
- Enhanced (Other): Clinics in the enhanced arm will receive core strategies along with enhanced strategies that involve more intensive training on depression treatment.
  Interventions: Other: Core Implementation Strategies; Other: Enhanced Implementation Strategies

INTERVENTIONS:
Other: Core Implementation Strategies — * Task Sharing/Revise Professional Roles
  * Distribute educational materials/Dynamic Training/Address Stigma
  * Clinician Implementation Team Meetings
  * Partner with CoCT DoH
  * Champion
  * Audit and Feedback
  * Stage Scale Up/Tailoring
Other: Enhanced Implementation Strategies — * Train the trainer
  * Ongoing supervision and consultation
  Arms: Enhanced

SUMMARY:
The goal of this clinical trial is to compare a core set and enhanced set of implementation strategies in increasing the reach of evidence-based treatments to patients with HIV and depression. The main questions it aims to answer are:

What proportion of patients start an evidence-based treatment for depression (reach)? What percentage of patients show clinical improvement in depression and what percentage attain viral undetectability within one year (effectiveness)?

Researchers will compare high and low reach clinics to further inform tailored implementation strategies for uptake and maintenance.

Clinics will be randomized into one of two study arms: core versus enhanced strategies. In both arms, core strategies will be utilized. Enhanced clinics will also receive more resource-intensive training.

ELIGIBILITY:
Inclusion Criteria for Clinics:

* Clinics are eligible if they provide HIV primary care via the City of Cape Town (CoCT) Department of Health
* Clinics will be assigned to the study upon notice of funding and before start up.

Inclusion Criteria for Patient-level Outcomes:

Although the unit of randomization is at the clinic level, the study will be looking at adult patient level data at each clinic. All patients engaged in care at one of the 10 primary care/HIV treatment clinics included in the study will be eligible to enroll if they:

* Are 18 years of age or older and
* Have a detectable HIV viral load (operationalized as the lower limit of detection on the standard test is used at the local clinic).
* Screen in for depression on the PHq-9 (score of 10 or above).

Exclusion Criteria:

-Children below the age of 18 will not be included in the proposed study for adults.

Inclusion Criteria for Qualitative data:

* For the qualitative data which involve interviewing clinic staff (specifically, nurses, physicians, clinic managers, or other involved in implementation) and patients, individuals will be eligible to participate if they are:
* employees (occupying the pre-specified roles) or patients (who met eligibility criteria for the implementation phase, regardless of whether or not they choose to enroll in the implementation phase) of a clinic that was randomized to the experimental condition.
* Clinic staff will be 18 years and older

Exclusion Criteria for Qualitative data:

- Children less than 18 will not be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2029-01-20 (Estimated); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Reach of depression treatment | 1 year
  Proportion of patients who start an evidence-based treatment for depression

SECONDARY OUTCOMES:
Depression | 1 year
  Percentage of patients, after one year, who are considered depression treatment responders (categorized as a responder if they achieve 50% reduction in symptoms on the PHQ-9 or if they no longer meet clinical criteria for depression).
Viral undetectability | 1 year
  Percentage of patients who attain an undetectable HIV RNA viral load across the two arms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
following NIH rules
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: This really depends on if the study will be reinstated
Access Criteria: This really depends on if the study will be reinstated

REFERENCES:
- [Background] Everitt-Penhale B, Kagee A, Magidson JF, Joska J, Safren SA, O'Cleirigh C, Witten J, Lee JS, Andersen LS. 'I went back to being myself': acceptability of a culturally adapted task-shifted cognitive-behavioural therapy (CBT) treatment for depression (Ziphamandla) for South African HIV care settings. Psychol Health Med. 2019 Jul;24(6):680-690. doi: 10.1080/13548506.2019.1566624. Epub 2019 Jan 17. PMID 30652921
- [Background] Safren SA, Bedoya CA, O'Cleirigh C, Biello KB, Pinkston MM, Stein MD, Traeger L, Kojic E, Robbins GK, Lerner JA, Herman DS, Mimiaga MJ, Mayer KH. Cognitive behavioural therapy for adherence and depression in patients with HIV: a three-arm randomised controlled trial. Lancet HIV. 2016 Nov;3(11):e529-e538. doi: 10.1016/S2352-3018(16)30053-4. Epub 2016 Sep 19. PMID 27658881
- [Background] Safren SA, O'Cleirigh C, Andersen LS, Magidson JF, Lee JS, Bainter SA, Musinguzi N, Simoni J, Kagee A, Joska JA. Treating depression and improving adherence in HIV care with task-shared cognitive behavioural therapy in Khayelitsha, South Africa: a randomized controlled trial. J Int AIDS Soc. 2021 Oct;24(10):e25823. doi: 10.1002/jia2.25823. PMID 34708929
- [Background] Safren SA, O'Cleirigh C, Tan JY, Raminani SR, Reilly LC, Otto MW, Mayer KH. A randomized controlled trial of cognitive behavioral therapy for adherence and depression (CBT-AD) in HIV-infected individuals. Health Psychol. 2009 Jan;28(1):1-10. doi: 10.1037/a0012715. PMID 19210012